CLINICAL TRIAL: NCT00096772
Title: Collection and Use of Blood For Genetic and Other Related Analyses (The GENOMICS Protocol)
Brief Title: Collection of Blood Samples From HIV Infected People
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPCRA 066; 10052 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2004-11-15; First posted 2004-11-16 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: HIV Infections
Keywords: Genetic Testing; Genomics; Human Genetic Factors
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Whole blood

SUMMARY:
The purpose of this study is to collect blood samples from HIV infected individuals for use in future genetic studies.

DETAILED DESCRIPTION:
Genetic differences among people with HIV may account for differences in disease progression and response to antiretroviral therapy. The Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA) was created to conduct studies in HIV infected communities and particularly in people of color, women, and injection drug users. This study will collect whole blood samples from HIV infected individuals. The samples will be used in future CPCRA studies comparing human genetic factors with clinical data from other CPCRA studies.

ELIGIBILITY:
Inclusion Criteria:

* Presently participating, previously participated in, or has given informed consent for participation in a qualifying CPCRA clinical trial
* Signed informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be selected from those who have given informed consent for participation in a qualifying CPCRA clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 2502 (Actual)
Dates: Start 2005-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Uy, MD, Study Chair — AIDS Research Alliance Chicago (ARAC), University of Illinois at Chicago
Locations (83):
- United States (83):
  - Dr. M. Estes Med. Practice CRS, Mill Valley, California
  - Dr. Robert Scott Med. Practice CRS, Oakland, California
  - East Bay AIDS Ctr. CRS, Oakland, California
  - Dr. Shawn Hassler Med. Practice CRS, San Francisco, California
  - Positive Health Program Clinic (San Francisco Gen. Hosp.) CRS, San Francisco, California
  - Dr. Virginia Cafaro Med. Practice CRS, San Francisco, California
  - Dr. William Owen Med. Practice CRS, San Francisco, California
  - Castro-Mission Health Ctr. CRS, San Francisco, California
  - St. Mary's Med. Ctr. of San Francisco CRS, San Francisco, California
  - San Francisco VAMC, Infectious Diseases Clinic CRS, San Francisco, California
  - UCSF PHP, Gen. Internal Medicine Practice CRS, San Francisco, California
  - Beacon Clinic at Boulder CRS, Boulder, Colorado
  - Denver Infectious Diseases Consultants CRS, Denver, Colorado
  - Kaiser Permanente of Denver CRS, Denver, Colorado
  - Univ. of Colorado Health Science Ctr. CRS, Denver, Colorado
  - Denver Public Health CRS - INSIGHT, Denver, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Eastside Family Health Ctr. CRS, Denver, Colorado
  - APEX Family Medicine CRS, Denver, Colorado
  - South Denver Infectious Diseases Specialists, Accord Med. Ctr. CRS, Denver, Colorado
  - Western Infectious Disease Consultants CRS, Wheat Ridge, Colorado
  - Yale Univ. School of Medicine, NE ProACT - New Haven CRS, New Haven, Connecticut
  - Georgetown Wellness Clinic, Georgetown, Delaware
  - Christiana Care Health Services HIV Program CRS, Wilmington, Delaware
  - Washington DC VAMC, Washington Regional AIDS Program, Infectious Diseases CRS, Washington D.C., District of Columbia
  - Klein & Slotten Medical Associates CRS, Chicago, Illinois
  - Univ. of Illinois Family Ctr. for Infectious Disease CRS, Chicago, Illinois
  - Lakeshore Infectious Disease Associates CRS, Chicago, Illinois
  - North Side Family Medicine CRS, Chicago, Illinois
  - Earl K. Long Med. Ctr., LSU - Mid City EIC Clinic CRS, Baton Rouge, Louisiana
  - James Osterberger, MD (Private Med. Practice) CRS, Baton Rouge, Louisiana
  - Med. Ctr. of Louisiana at New Orleans, HIV Outpatient Clinics CRS, New Orleans, Louisiana
  - Tulane University Health Sciences Center, Louisiana Community AIDS Research Program(LaCARP) CRS, New Orleans, Louisiana
  - New Orleans VAMC CRS, New Orleans, Louisiana
  - CRI-Boston CRS, Boston, Massachusetts
  - CRI-Springfield CRS, Springfield, Massachusetts
  - Harper Hosp., Detroit CRS, Detroit, Michigan
  - Wayne State Univ. CRS, Detroit, Michigan
  - Wayne State Univ. INSIGHT CRS, Detroit, Michigan
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Henry Ford Hosp., Div. of Infectious Disease INSIGHT CRS, Detroit, Michigan
  - Detroit Community Health Connection, Inc. CRS, Detroit, Michigan
  - Univ. of Mississippi Med. Ctr., Div. of Infectious Diseases CRS, Jackson, Michigan
  - Michigan State Univ., Infectious Disease Clinic CRS, Lansing, Michigan
  - Cooper Hospital/Univ. Med. Ctr., The Cooper Early Intervention Program (EIP) CRS, Camden, New Jersey
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - ID Care Inc. - Hillsborough CRS, Hillsborough, New Jersey
  - Jersey Shore Univ. Med. Ctr. CRS, Neptune City, New Jersey
  - Cathedral Healthcare System, St. Michael's Med. Ctr. CRS, Newark, New Jersey
  - New Jersey Community Research Initiative, Jeffrey Bomser Clinic CRS, Newark, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey CRS, Paterson, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey, Paterson, New Jersey
  - Raritan Bay Med. Ctr., Perth Amboy Division CRS, Perth Amboy, New Jersey
  - ID Care - Randolph CRS, Randolph Township, New Jersey
  - Infectious Disease Specialists of N.J., North Jersey Community Research Initiative CRS, Union, New Jersey
  - The Early Intervention Program at Kennedy Hosp. CRS, Voorhees Township, New Jersey
  - St. Vincent Hosp. & Med. Ctr. CRS, New York, New York
  - Harlem Hospital Ctr./Columbia University CRS (Gordin CTU), New York, New York
  - Harlem Hosp. Ctr., Outpatient Clinics (New York) CRS, New York, New York
  - Bronx- Lebanon Hospital Center Clinical Research Site (BLHC CRS), The Bronx, New York
  - Bronx-Lebanon Hosp. Ctr. CRS, The Bronx, New York
  - Montefiore Med. Ctr., AIDS Ctr. CRS, The Bronx, New York
  - Multnomah County Health Dept., HIV Health Services Ctr. CRS, Portland, Oregon
  - Legacy Clinic Good Samaritan CRS, Portland, Oregon
  - The Research & Education Group-Portland CRS, Portland, Oregon
  - Providence Portland Med. Ctr., Ambulatory Care and Education Ctr. CRS, Portland, Oregon
  - Kaiser Immune Deficiency Clinic of Portland CRS, Portland, Oregon
  - Legacy Clinic Emanuel CRS, Portland, Oregon
  - Legacy Clinic Northeast CRS, Portland, Oregon
  - Oregon Health & Sciences Univ. Internal Medicine (L-475) CRS, Portland, Oregon
  - Temple Univ. School of Medicine CRS, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Thomas St. Clinic CRS, Houston, Texas
  - Houston AIDS Research Team CRS, Houston, Texas
  - Michael E. DeBakey VAMC CRS, Houston, Texas
  - Thomas Street Clinic CRS, Houston, Texas
  - MediCorp, Infectious Disease Associates CRS, Fredericksburg, Virginia
  - Petersburg Health Care Alliance CRS, Petersburg, Virginia
  - Vernon Harris East End Community Health Ctr. CRS, Richmond, Virginia
  - CrossOver Health Ctr. CRS, Richmond, Virginia
  - South Richmond Health Care Ctr. CRS, Richmond, Virginia
  - Hunter Holmes McGuire VAMC CRS, Richmond, Virginia
  - VCU Health Systems, Infectious Disease Clinic CRS, Richmond, Virginia
  - Virginia Commonwealth Univ. Medical Ctr. CRS, Richmond, Virginia

REFERENCES:
- [Background] Anastassopoulou CG, Kostrikis LG. The impact of human allelic variation on HIV-1 disease. Curr HIV Res. 2003 Apr;1(2):185-203. doi: 10.2174/1570162033485311. PMID 15043202
- [Background] O'Brien SJ, Nelson GW. Human genes that limit AIDS. Nat Genet. 2004 Jun;36(6):565-74. doi: 10.1038/ng1369. PMID 15167933
- [Background] Telenti A. The genetic cohorts: facing the new challenges in infectious diseases. The HIV model. Enferm Infecc Microbiol Clin. 2004 Jun-Jul;22(6):337-41. doi: 10.1016/s0213-005x(04)73106-7. PMID 15228901